CLINICAL TRIAL: NCT03692351
Title: Osteolysis Development Over Time Around Uncemented Titanium Fiber Mesh Cups With or Without Screw Holes
Brief Title: Osteolysis Development Around Uncemented Cups With or Without Screw Holes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Per-Erik Johanson, Researcher, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protesteam_Trilogy
Record Dates: First submitted 2018-08-20; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Arthroplasty Complications
Keywords: uncemented hip arthroplasty; osteolysis; polyethylene wear; implant design
MeSH Terms: conditions — Osteolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cup with screw holes (Active Comparator): Uncemented Trilogy cup (Zimmer, Warzaw, IN, US), screw fixation (2 or 3 screws)
  Interventions: Device: Uncemented acetabular cup with screw holes
- Cup without screw holes (Experimental): Uncemented Trilogy cup (Zimmer, Warzaw, IN, US) without screw holes, press-fit fixation
  Interventions: Device: Uncemented acetabular cup without screw holes

INTERVENTIONS:
Device: Uncemented acetabular cup with screw holes
  Arms: Cup with screw holes
Device: Uncemented acetabular cup without screw holes
  Arms: Cup without screw holes

SUMMARY:
In order to investigate the role of acetabular cup screw holes for the transport of osteolysis-inducing particles in a total hip arthroplasty articulation, the investigators compare the amount of bone loss around acetabular cups with and without holes. Bone loss is measured with computed tomography at 7 years and 15 - 18 years of follow-up.

DETAILED DESCRIPTION:
Particles generated by wear and corrosion within an artificial hip articulation can cause biologically mediated bone loss in the surrounding pelvis. Particles can be found within immunologically active cells inside bone lesions. Holes intended for screw fixation in uncemented acetabular cups are believed to be a main route for these particles from the articulation into the pelvic bone. Using pressfit, screws are not always necessary for a successful fixation of an uncemented cup. The investigator's hypothesis is that a pressfit fixated cup without screw holes will display a decreased amount of periacetabular osteolysis compared to a cup with screw holes. Therefore, 95 hips (90 patients) were randomized to receive either pressfit cups without screw holes or the same type of cup with screw holes. The occurence and size of periacetabular osteolysis will be compared between the two groups. In addition, since the patients will have a computed tomography examination at 7 years and between 15 and 18 years the investigator will also analyze development of periacetabular osteolysis over time. The different cups were paired with three different types of femoral stems. Also, articulation wear and cup and stem fixation will be analyzed using radiostereometry.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary osteoarthritis

Exclusion Criteria:

* Inflammatory osteoarthritis, hip joint infection

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 1994-06-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Periacetabular osteolysis frequency change between 7 and 18 years | Change between 7 to 18 years after surgery
  Frequency of osteolysis (%) measured with computed tomography
Periacetabular osteolysis size change between 7 and 18 years | Change between 7 to 18 years after surgery
  Size of periacetabular osteolysis (cm3) masured with computed tomography

SECONDARY OUTCOMES:
Cup fixation (translation) | 18 years postoperatively
  Cup translation (mm/year) measured with radiostereometry, calculated from multiple measurements during the study period
Cup fixation (rotation) | 18 years postoperatively
  Cup rotation (degrees/year) measured with radiostereometry, calculated from multiple measurements during the study period
Polyethylene wear | 18 years postoperatively
  Polyethylene wear (mm/year) measured with radiostereometry, calculated from multiple measurements during the study period

IPD SHARING:
Plan to Share IPD: No